CLINICAL TRIAL: NCT07154953
Title: Serum Surfactant Protein-D and Inflammatory Biomarkers as Predictors of Disease Severity in Hospitalized Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Serum Surfactant Protein-D as Predictor of Disease Severity in Hospitalized COPD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mostafa Ahmed Mohamed, Principal Investigator, Assiut University
Other Study IDs: SP-D in COPD
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with acute COPD exacerbation admitted to ICU: * Adults ≥40 years diagnosed with COPD based on prior diagnosis or spirometry if available.
  * Admission for acute exacerbation (AECOPD) in Respiratory ICU.
  Interventions: Diagnostic Test: Serum Surfactant Protein-D
- patients with COPD admitted to ward settings: * Adults ≥40 years diagnosed with COPD based on prior diagnosis or spirometry if available.
  * Admission for acute exacerbation (AECOPD) in ward .
  Interventions: Diagnostic Test: Serum Surfactant Protein-D

INTERVENTIONS:
Diagnostic Test: Serum Surfactant Protein-D — Several studies support the use of SP-D as a marker of systemic inflammation and lung tissue damage in COPD.Measuring serum SP-D could provide a valuable tool for early detection, monitoring progression, and personalizing management of COPD patients.Surfactant protein D (SP D) as a prognostic biomarker needs further studies to validate its clinical applicability

SUMMARY:
evaluation of the serum levels of surfactant protein-D (SP-D), C-reactive protein (CRP), fibrinogen, and peripheral blood neutrophilic and eosinophilic counts in patients with COPD correlation of these biomarkers with clinical, functional, and radiological parameters

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic progressive inflammatory disease of the airways and lungs, mainly caused by cigarette smoking and environmental exposures .It is characterized by airflow limitation that is not fully reversible, with exacerbations and systemic manifestations.

In COPD, there is a significant immune dysregulation, involving both innate and adaptive immune responses.Surfactant Protein D (SP-D) is a lung-specific collectin, produced primarily by alveolar type II cells and Clara cells.SP-D plays a key role in the innate immune defense of the lungs, particularly in modulating inflammation, enhancing phagocytosis, and neutralizing pathogens.

In COPD, the epithelial barrier is compromised, leading to increased leakage of SP-D from the lungs into the bloodstream.As a result, serum levels of SP-D are elevated in COPD patients, and this elevation is positively associated with disease severity and exacerbation frequency.

.SP-D has been proposed as a non-invasive biomarker for COPD severity, progression, and response to therapy.Several studies support the use of SP-D as a marker of systemic inflammation and lung tissue damage in COPD.Measuring serum SP-D could provide a valuable tool for early detection, monitoring progression, and personalizing management of COPD patients.Surfactant protein D (SP D) as a prognostic biomarker needs further studies to validate its clinical applicability.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥40 years diagnosed with COPD based on prior diagnosis or spirometry if available.
* Admission for acute exacerbation (AECOPD) in ward or Respiratory ICU.

Exclusion Criteria:

* Active pulmonary infection unrelated to COPD (e.g. tuberculosis, fungal infections)
* Other chronic lung diseases such as asthma, interstitial lung disease, or lung cancer
* Use of systemic corticosteroids for conditions other than COPD exacerbation

Ages: 40 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults ≥40 years diagnosed with COPD based on prior diagnosis or spirometry if available.
  Admission for acute exacerbation (AECOPD) in ward or Respiratory ICU.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of serum SP-D levels | baseline
  To evaluate serum SP-D levels in patients with acute COPD exacerbation admitted to ICU and ward settings

SECONDARY OUTCOMES:
• Correlation of SP-D with: o Systemic inflammatory markers (CRP, fibrinogen, eosinophils, NLR) o Symptom burden and dyspnea scores (CAT, mMRC) o Prognostic scores (DECAF, APACHE II) o Basic CT chest findings | baseline
  • Correlate SP-D with:
  * Systemic inflammatory markers (CRP, fibrinogen, eosinophils, NLR)
  * Symptom burden and dyspnea scores (CAT, mMRC)
  * Prognostic scores (DECAF, APACHE II)
  * Basic CT chest findings

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ahmed Abdelhafeez, Professor, Principal Investigator — Assiut University; HA Abdelhafeez, Professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zemans RL, Jacobson S, Keene J, Kechris K, Miller BE, Tal-Singer R, Bowler RP. Multiple biomarkers predict disease severity, progression and mortality in COPD. Respir Res. 2017 Jun 13;18(1):117. doi: 10.1186/s12931-017-0597-7. PMID 28610627
- [Background] He X, Ji J, Zheng D, Luo Z, Luo L, Guo L. Serum surfactant protein D as a significant biomarker for predicting occurrence, progression, acute exacerbation, and mortality in interstitial lung disease: a systematic review and meta-analysis. Front Immunol. 2025 Feb 14;16:1450798. doi: 10.3389/fimmu.2025.1450798. eCollection 2025. PMID 40028331